CLINICAL TRIAL: NCT04829097
Title: A Prospective Multicenter Randomized Controlled Clinical Trial of Neoadjuvant Temozolomide Combined With Simultaneous Increased Intensity-modulated Radiotherapy in the Treatment of Glioblastoma
Brief Title: Neoadjuvant Temozolomide Combined With Simultaneous IMRT for Treatment of Glioblastoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Yang Yang, Professor of medicine, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-307-02
Record Dates: First submitted 2021-03-25; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIB-IMRT (Experimental): 1. New auxiliary TMZ period: oral TMZ 75mg/m2, qd, continued until the beginning of radiotherapy. 2. Concurrent radiotherapy and chemotherapy period: 4 weeks in total. Prior to treatment, radiotherapy positioning and planning were established, using SIB-IMRT technology, the irradiation range, the tumor residual area 60Gy/20f/4w, the tumor bed area 40Gy/20f/4w, 1 time/d, 5 times/w. During radiotherapy, TMZ will continue to be administered orally simultaneously, the specific dose: TMZ 75mg/m2 qd, until 42 days. 3. Intermediate rest period: 4 weeks in total. ;4. TMZ adjuvant chemotherapy period: 6 to 12 months in total. Cycle 1: TMZ 150mg/m2, d1-5, q28d; if the patient can tolerate it, cycles 2-12: TMZ 200mg/m2, d1-5, q28d; after cycles 3, 6, 9, and 12 of adjuvant chemotherapy Head functional magnetic resonance examination was performed to assess the size of residual lesions and edema.
  Interventions: Combination Product: Temozolomide
- CRT (Active Comparator): 1. Concurrent radiotherapy and chemotherapy period: 6 weeks in total. Radiotherapy positioning and planning before treatment, using CRT technology, irradiation range, tumor bed area, 60Gy/30f/6w, 1 time/d, 5 times/w, simultaneous TMZ oral administration on the first day of radiotherapy, specific dose: TMZ 75mg/m2 qd for 42 consecutive days; head functional magnetic resonance imaging was performed at the end of radiotherapy to assess the size of residual lesions and edema. 2. Intermediate rest period: 4 weeks in total. The patient will go to the hospital to recheck blood routine every week;3. TMZ adjuvant chemotherapy period: 6 to 12 months in total. Cycle 1: TMZ 150mg/m2, d1-5, q28d; if the patient can tolerate it, cycles 2-12: TMZ 200mg/m2, d1-5, q28d; head functional magnetic resonance imaging was performed after adjuvant chemotherapy in cycles 3, 6, 9, and 12 to assess the size of residual lesions and edema.
  Interventions: Combination Product: Temozolomide

INTERVENTIONS:
Combination Product: Temozolomide — The patient received neoadjuvant temozolomide combined with simultaneous increase in intensity-modulated radiotherapy. According to data from previous clinical trials, neoadjuvant temozolomide combined with concurrently increased intensity-modulated radiotherapy PFS for 13.7 months.
  Other Names: Intensity-Modulated Radiotherapy

SUMMARY:
This study is a prospective, multi-center, randomized controlled clinical study. Indications: Glioblastoma diagnosed after surgery (WHO grade IV). The patient received conventional postoperative concurrent radiotherapy and chemotherapy, or neoadjuvant temozolomide combined with concurrent increased intensity-modulated radiotherapy. According to data from previous clinical trials, conventional doses of concurrent radiotherapy and chemotherapy PFS 6.9 months neoadjuvant temozolomide combined with concurrently increased intensity-modulated radiotherapy PFS 13.7 months, an estimated 20% leakage rate, and a total sample size of 80 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 70 years old
* A patient with high-grade (WHO grade IV) glioma diagnosed pathologically
* ECOG score ≤ 3 points
* The expected survival time is greater than 3 months
* Patients undergoing surgery for the first time
* Patients who have not received radiotherapy at the treatment site in the past
* The following hematological indicators need to be met Neutrophil count ≥1.5×109/L Hemoglobin ≥9g/dL Platelet count ≥70×109/L
* The following biochemical indicators need to be met Total bilirubin≤1.5×upper limit of normal (ULN) AST and ALT<1.5×ULN Creatinine clearance rate ≥60ml/min
* Patients of childbearing age need to take appropriate protective measures (contraception or other methods of birth control) before enrollment and during the trial
* The signed informed consent form
* Ability to follow research protocols and follow-up procedures

Exclusion Criteria:

* Patients with recurrent glioma who have previously undergone surgery or radiotherapy and chemotherapy
* Glioma of the spinal cord
* ECOG score> 3 points
* Severe mental symptoms; uncontrollable status epilepticus
* Patients with malignant tumors in other parts
* The patient has an active bacterial, viral or fungal infection (≥ Grade 2 NCI-CTC, 4th edition)
* The patient has severe liver and kidney dysfunction, HIV infection, HCV infection, uncontrollable coronary artery disease or asthma, uncontrollable cerebrovascular disease or other diseases that the researcher thinks cannot be included in the group
* Pregnant and lactating women. Women of childbearing age must have a negative pregnancy test within 7 days before joining the group
* Drug abuse, clinical, psychological or social factors affect informed consent or research implementation
* Any uncertain factors that affect the safety or compliance of patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Two years after all treatments are over
  RANO criteria: evaluate the therapeutic effect of glioma through MRI and clinical manifestations.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China